CLINICAL TRIAL: NCT05508607
Title: Precision Antimicrobial STewardship for Clostridioides DIfficile Prevention
Acronym: PASTCDI
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1051390
Record Dates: First submitted 2020-05-27; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: CDI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Implementation
- Post-Implementation
  Interventions: Other: CDI-risk Classification Tool

INTERVENTIONS:
Other: CDI-risk Classification Tool — This tool will focus a bundle of antimicrobial stewardship (AMS) CDI prevention recommendations on high-risk patients.
  Groups: Post-Implementation

SUMMARY:
To decrease CDI incidence by implementing an electronic health record-integrated CDI-risk classification tool for Clostridioides difficile infection (CDI) to focus a bundle of antimicrobial stewardship (AMS) CDI prevention recommendations on high-risk patients.

DETAILED DESCRIPTION:
This study aims to use a pre/post implementation design to evaluate the use of a novel risk classification tool to improve existing methods of identifying patients eligible for routine antimicrobial stewardship (AMS) care processes targeting reduction of Clostridioides difficile infection (CDI). Antimicrobial stewardship is an established, evidence-based quality improvement program that is required by The Joint Commission and a condition of participation by the Centers for Medicare and Medicaid. AMS processes of care are evidence based, supported by published research demonstrating outcomes benefits, are recommended by national guidelines and are not investigational. Treatment decisions remain at the discretion of clinicians and patients

ELIGIBILITY:
Inclusion Criteria:

* adult acute care patients identified as high-CDI risk by the CDI risk classification tool. This sub-group represents approximately 6% of all acute care admissions

Exclusion Criteria:

* Behavioral health units
* Inpatient rehabilitation units
* Labor and Delivery units
* Same day surgery and observation units

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our goal is to study the all adults admitted to any of the 22 Intermountain Healthcare network acute care hospitals who are classified as high risk for CDI by the risk classification tool. In this pre-post design study, we will identify two cohorts, the first representing a two-year cohort prior to implementation of the risk classification-enhanced AMS process and the second a post-implementation cohort representing one-year after implementation. These cohorts will be identified retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 13319 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Per-Admission Rate | 30 days after discharge
  per-admission rate of hospital-associated CDI, defined as: positive toxin B by enzyme-linked immunoassay or polymerase chain reaction test at least 72 hours after admission

SECONDARY OUTCOMES:
Total Antibiotic Usage | through study completion, an average of 1 year
High-Risk Antibiotic Usage | through study completion, an average of 1 year
Proton Pump Inhibitor Therapy Administered | through study completion, an average of 1 year
Total Variable Cost per Admission | through study completion, an average of 1 year
Hospital Length of Stay | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No